CLINICAL TRIAL: NCT07144137
Title: A Non-Interventional Study Observing Short-Term Progression in Geographic Atrophy (GA) Secondary to Age-Related Macular Degeneration (AMD)
Brief Title: A Non-Interventional Study Observing Short-Term Progression in Geographic Atrophy (GA)
Acronym: Pre-GAIN
Status: Recruiting | Type: Observational
Sponsor: Complement Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: IGS02
Record Dates: First submitted 2025-08-20; First posted 2025-08-27 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Geographic Atrophy Secondary to Age-related Macular Degeneration
Keywords: GA; AMD; Geographic atrophy; Dry AMD; Age-related macular degeneration
MeSH Terms: conditions — Geographic Atrophy; Macular Degeneration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a non-interventional, observational study to provide insights into the short-term progression of GA secondary to AMD in participants aged ≥55 years.

This is a multi-center, non-interventional, observational study which aims to identify participants who have progressive GA to allow quantification of structural and functional parameters that characterize the progression of GA, and to investigate whether these correlate with genetic or lifestyle factors.

ELIGIBILITY:
Inclusion:

1. Participants must be aged ≥55 years, at the time of signing the informed consent at the screening visit.
2. Participants with bilateral GA secondary to AMD as confirmed by the Central Reading Center using FAF and/or OCT images with at least 1 eye having a total GA lesion area must be between 1.25 mm2 and 17.5 mm2 inclusive, determined by FAF images taken at the screening visit.
3. Best-corrected visual acuity (BCVA) in both eyes should be sufficient to ensure navigational vision (defined as 20/400 or better for purposes of this study).
4. BCVA between 20 and 75 letters and LLVA>0 letters using an ETDRS chart.
5. Mean retinal sensitivity as measured by microperimetry using the study grid must be equal to or greater than 5 dB.
6. Able and willing to provide signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol, and in the opinion of the investigator, is able to perform all study assessments.

Exclusion criteria:

1. Macular atrophy secondary to any condition other than AMD in the study eye.
2. Any pathology of the macula other than GA secondary to AMD and other changes consistent with early, intermediate or atrophic AMD in the study eye.
3. Evidence of prior or current Choroidal Neovascularization (CNV), also known as wet-AMD, in either eye.
4. Atrophic retinal disease of causality other than AMD including monogenetic macular dystrophies (incorporating pattern dystrophy), myopia-related maculopathy and Stargardt disease in the study eye.
5. A history of vitrectomy in the study eye.
6. Any prior treatment for AMD or any prior intravitreal treatment for any indication in the study eye, except oral supplements of vitamins and minerals such as the age-related eye disease study (AREDS) formula.
7. Any intraocular surgery (except cataract surgery within 6 months of enrollment) or thermal laser within 3 months of screening, or any ophthalmic condition that may require surgery during the study.
8. Any macular laser, macular surgery or retinal surgery at any time point in the study eye.
9. Any ocular or periocular infection in the 12 weeks prior to screening.
10. History of uveitis or endophthalmitis in either eye.
11. Any sign of diabetic retinopathy in either eye, or HbA1c >8, in the 12 months prior to enrollment.
12. High myopia or hyperopia (≥6 diopter) in the study eye.
13. Uncontrolled IOP measurement of ≥25 mmHg for >1 month despite being on 2 or more ocular hypotensive agents, or IOP >21 mm Hg in the presence of C/D asymmetry of >0.3 per the reading center; or glaucomatous damage to the optic nerve or visual field.
14. Retinal disease other than AMD or other ocular disorders which may cause safety concerns per the judgment of the investigator; however, benign conditions of the vitreous or peripheral retina are not exclusionary (i.e., paving stone degeneration).
15. Any ophthalmologic condition that reduces the clarity of the media and that, in the opinion of the investigator interferes with ophthalmologic examination (e.g., cataract or corneal abnormalities) either at the time of enrollment or during the 2-year post dosing follow-up period; or prevents adequate imaging of the retina judged by the site or CRC.
16. Aphakia or absence of the posterior capsule. Previous violation of the posterior capsule is also excluded unless it occurred as a result of yttrium aluminum garnet (YAG) laser posterior capsulotomy in association with prior posterior chamber intraocular lens implantation and at least 60 days prior to baseline.
17. Medical or psychiatric conditions that, in the opinion of the investigator, make consistent follow-up over the treatment period unlikely, or in general a poor medical risk because of other systemic diseases or active uncontrolled infections, including but not limited to immunodeficiency state, autoimmune diseases, malignancy other than prostate or basal cell carcinoma, connective tissue disorders and collagen vascular disorders.
18. Participation in an interventional clinical study, or use of any experimental treatment for AMD or any investigational product within 6 months or 5 half-lives of the active ingredient (whichever is longer) prior to screening.
19. History of abnormal laboratory tests (e.g. hematology, serum chemistry, renal or liver function tests, or infectious disease screen) that in the opinion of the investigator is clinically significant at the time of enrollment and not suitable for study participation.
20. Hypersensitivity to medications used in (standard of care) study procedures.
21. Situations where, in the opinion of the investigator, the risk of harm to a participant outweighs any potential benefits from study participation (these could include participants with conditions such as brittle diabetes or advanced osteoporosis as examples).
22. History or current use of medications associated with macular changes, retinal dysfunction or optic nerve damage. These include but are not limited to the following prohibited concomitant medications:
23. Any previous gene or cell therapy (ophthalmic or systemic),
24. Chloroquine (where taken for >30 days cumulative across participant's lifetime), hydroxychloroquine, platinum containing medications, ethambutol, tamoxifen, pentosan, chronic use of phosphodiesterase inhibitors, and GLP-1 antagonists in the setting of a crowded optic disc.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female participants, aged ≥55 years, with GA secondary to AMD are considered the appropriate population. This represents the lower end of the age range for the population with GA secondary to AMD with appropriately advanced disease to enable the measurement of disease progression.
  Participants with bilateral GA are selected to minimize the risk of developing neovascular (wet) AMD during the study and to allow the collection of data and potential comparison of progression for 2 eyes for each participant.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2025-07-30 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Short-term GA Progression | Baseline, Month 3, Month 6
  To quantify the structural and functional parameters of short-term progression of geographic atrophy (GA) through clinical evaluation and investigations

SECONDARY OUTCOMES:
Further exploration of GA progression | Baseline, Month 3, Month 6
  To further explore selected potential correlates of structural and functional parameters of GA progression in greater depth

CONTACTS AND LOCATIONS:
Locations (1):
- Sierra Eye Associates, Reno, Nevada, United States

IPD SHARING:
Plan to Share IPD: No